CLINICAL TRIAL: NCT04031859
Title: The Effectiveness of a Risk Stratification Procedure for Thromboembolism Prophylaxis After Total Knee Replacement Surgeries
Brief Title: Risk Stratification Procedure for Thromboembolism Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Collaborators: Prince Sultan Military College of Health Sciences (Other); Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mariam Ahmad Alameri, Clinical Pharmacist, Clinical Pharmacist, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSMMC & KAAUH
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Total Knee Replacement Surgeries
Keywords: Total Knee Replacement; Venous thromboembolism (VTE); Risk Stratification
MeSH Terms: conditions — Venous Thromboembolism | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): In this group a VTE risk stratification procedure will be used
  Interventions: Drug: acetylsalicylic acid
- Group B (No Intervention): In this group a standard VTE risk stratification procedure will be used (Caprini VTE risk assessment tool)

INTERVENTIONS:
Drug: acetylsalicylic acid — It's a VTE risk stratification tool or procedure that will be used after total knee replacement (TKR) to help surgeons in choosing the tailored VTE prophylaxis according to patients' specific VTE risk, this tool will stratify the TKR-patient in one of three risk-groups: Low high risk who will be prescribed Aspirin upon hospital discharge as extended VTE prophylaxis post TKR surgery, or moderate high risk group who will be prescribed oral anti coagulant (like rivaroxaban) as extended prophylaxis, and the last group is very high risk group who will be prescribed parenteral anticoagulant ( like Enoxaparin) plus compression devices.
  Other Names: VTE risk stratification procedure
  Arms: Group A

SUMMARY:
The main objective for this study is validation for the proposed risk stratification tool, by evaluating the clinical outcomes for its use post TKR Surgeries. For this objective, the design that is used is Randomized Trial.

DETAILED DESCRIPTION:
All patients that will have total knee replacement, in a given period of time in both medical centers; Prince Sultan Military Medical City (PSMMC) and King Abd Allah University Hospital (KAAUH) in Princess Noura University, will be randomly separated into 2 groups; in the first group (A): Venous thromboembolism (VTE) risk stratification tool (which is prepared by a clinical pharmacist) will be applied to choose the tailored extended VTE prophylactic agent. While in the second group (B), the risk stratification tool will not be used, rather it will follow the routine hospital protocol for choosing the VTE prophylactic agent, which is Caprini: a standard validated model. Then each group of patients will be followed till 35 days post-operation, during which all VTE or bleeding events should be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients who are planned for elective TKR surgery (primary only).
2. Agreed to sign the Informed consent form (ICF).
3. Patients aged older than 18 years.

Exclusion Criteria:

1. Patients receiving anticoagulant for treatment.
2. Patients with a history of DVT or PE were excluded from the study due to the marked increase in the risk of recurrent VTE compared to the general risk of (7% vs. 0.1%); (Fahrni, 2015).
3. Patients with renal or hepatic failure, renal failure is defined as end-stage kidney disease (on dialysis); hepatic failure is defined as complete liver cirrhosis.
4. Pregnant woman.
5. Revision surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-07-14 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism (VTE) complications | 35 days post total Knee Replacement surgery
  Deep vein thrombosis, pulmonary embolism, sudden death
Bleeding events | 35 days post total Knee Replacement surgery
  Major or minor bleeding will be recorded

SECONDARY OUTCOMES:
Surgical site infection | 35 days post total Knee Replacement surgery
  Surgical site infection post operation

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Alameri, MSC, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Prince Sultan Medical Military City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alameri MA, Syed Sulaiman SA, Ashour AM, Al-Saati MF. Venous thromboembolism prevention protocol for adapting prophylaxis recommendations to the potential risk post total knee replacement: a randomized controlled trial. Pharm Pract (Granada). 2020 Jul-Sep;18(3):2025. doi: 10.18549/PharmPract.2020.3.2025. Epub 2020 Sep 22. PMID 33029262